CLINICAL TRIAL: NCT07392320
Title: A Randomized, Open-Label, Phase II Clinical Study Comparing Immunotherapy Combined With Induction Chemotherapy Followed by Concurrent Chemoradiotherapy and Immunotherapy Maintenance Versus Capecitabine Maintenance in Locally Advanced High-Risk Nasopharyngeal Carcinoma
Brief Title: A Phase II Trial Comparing Immunotherapy Versus Capecitabine Maintenance After Chemo-chemoradiotherapy for High-risk Nasopharyngeal Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Pei-Yu Huang, Principal Investigator, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-FXY-476
Record Dates: First submitted 2026-01-26; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Nasopharangeal Cancer
Keywords: high-risk locally advanced nasopharyngeal carcinoma
MeSH Terms: interventions — spartalizumab; Capecitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adjuvant immunotherapy arm (Experimental): Adjuvant PD-1 monoclonal antibody maintenance
  Interventions: Drug: TP+PD1+CCRT; Drug: PD-1 Monoclonal Antibody
- Adjuvant chemotherapy arm (Experimental): Adjuvant capecitabine maintenance
  Interventions: Drug: TP+PD1+CCRT; Drug: Capecitabine

INTERVENTIONS:
Drug: TP+PD1+CCRT — Induction Chemoimmunotherapy (3 cycles, Q3W):
  Induction chemotherapy consisted of three cycles of docetaxel (75 mg/m², day 1), cisplatin (75 mg/m², day 1), and penpulimab (200 mg, day 1), administered every 3 weeks.
  Concurrent Chemotherapy (3 weeks post-induction, 2 cycles, Q3W):
  concurrent cisplatin 100mg/m2 every 21days for two cycles during Intensity modulated-radiotherapy (IMRT)
Drug: PD-1 Monoclonal Antibody — Penpulimab 200 mg every 3 weeks for 8 cycles
  Arms: Adjuvant immunotherapy arm
Drug: Capecitabine — Capecitabine 1000 mg/m² BID, days 1-14, for 8 cycles.
  Arms: Adjuvant chemotherapy arm

SUMMARY:
In this study, the investigators designed a randomized, open-label, phase II clinical trial for high-risk locally advanced nasopharyngeal carcinoma (T4 or N3 or EBV DNA ≥1500 copies/ml, AJCC 9th edition) that is sensitive to chemotherapy and PD-1 monoclonal antibody therapy. The trial compares sequential treatment with the TP regimen combined with PD-1 monoclonal antibody followed by concurrent chemoradiotherapy and PD-1 maintenance therapy versus capecitabine maintenance therapy. The aim is to provide high-quality clinical evidence for optimizing the treatment strategy for high-risk locally advanced nasopharyngeal carcinoma.

DETAILED DESCRIPTION:
For high-risk locally advanced nasopharyngeal carcinoma, it remains essential to explore more effective treatment strategies and regimens. In the era of immunotherapy, the introduction of PD-1 monoclonal antibodies has provided significant survival benefits to patients with locally advanced nasopharyngeal carcinoma. However, different modes of intervention still warrant further exploration, and additional clinical evidence is needed for validation.

In this study, the investigators designed a randomized, open-label, phase II clinical trial focusing on high-risk locally advanced nasopharyngeal carcinoma (defined as T4 or N3 or EBV DNA ≥1500 copies/ml according to AJCC 9th edition) that is sensitive to chemotherapy and PD-1 monoclonal antibody therapy. The trial compares the sequential approach of TP regimen combined with PD-1 monoclonal antibody followed by concurrent chemoradiotherapy and PD-1 maintenance therapy versus maintenance therapy with capecitabine. The study aims to provide high-quality clinical evidence to optimize treatment strategies for high-risk locally advanced nasopharyngeal carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary participation and written informed consent must be signed.
* Age between 18 and 70 years, male or non-pregnant female.
* Pathologically confirmed nasopharyngeal non-keratinizing carcinoma (differentiated or undifferentiated type, i.e., WHO type II or type III).
* Stage III disease (AJCC 9th edition staging) or pre-treatment plasma Epstein-Barr virus DNA (EBV DNA) ≥ 1500 copies/ml.
* Efficacy after 3 cycles of induction immunochemotherapy assessed as complete response (CR) or partial response (PR) by nasopharyngoscopy and contrast-enhanced MRI of the nasopharynx and neck.
* ECOG performance status score of 0 or 1.
* Adequate hematological function: Hemoglobin (HGB)≥90g/L, White Blood Cell (WBC) ≥ 4.010^9/L, and Platele (PLT) ≥10010^9/L.
* Adequate hepatic function: ALT and AST≤2.5Upper Limit of Normal (ULN), total bilirubin ≤2.0ULN, and serum albumin≥30g/L.
* Adequate renal function: Serum creatinine ≤ 1.5*ULN or calculated creatinine clearance (CrCl) ≥ 60 mL/min (using the Cockcroft-Gault formula).
* International Normalized Ratio (INR) and Activated Partial Thromboplastin Time (APTT) ≤ 1.5 *ULN (unless the subject is receiving anticoagulant therapy and the coagulation parameters (PT/INR and APTT) are within the expected therapeutic range for the anticoagulant at the time of screening).

Exclusion Criteria:

* Patients with recurrent or distant metastatic nasopharyngeal carcinoma.
* Pathological diagnosis of keratinizing squamous cell carcinoma (WHO Type I).
* Patients who have previously received radiotherapy or systemic chemotherapy.
* Women who are pregnant or breastfeeding, or individuals of childbearing potential who are not using effective contraception.
* HIV positive.
* History of other malignancies (except for cured basal cell carcinoma or cervical carcinoma in situ).
* Patients who have previously received immune checkpoint inhibitors (e.g., CTLA-4, PD-1, PD-L1 inhibitors).
* Patients with immunodeficiency diseases or a history of organ transplantation.
* History of autoimmune diseases, including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis.
* Patients who have received high-dose glucocorticoids, anticancer monoclonal antibodies, or other immunosuppressive therapy within 4 weeks.
* Patients with significantly impaired cardiac, hepatic, pulmonary, renal, or bone marrow function.
* Patients with severe, uncontrolled medical conditions or infections.
* Concurrent use of other investigational drugs or participation in another clinical trial.
* Refusal or inability to sign the informed consent form for trial participation.
* Patients with other contraindications to the treatment.
* Patients with personality or psychiatric disorders, or those lacking or with limited legal capacity.
* Patients who are hepatitis B surface antigen (HBsAg) positive with peripheral blood hepatitis B virus DNA (HBV DNA) ≥ 1000 copies/ml. Patients who are HBsAg positive but have HBV DNA < 1000 copies/ml are eligible if the investigator determines that their chronic hepatitis B is stable and does not pose an increased risk.
* Patients with a positive HCV antibody test result, unless the polymerase chain reaction (PCR) test for HCV RNA is negative.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2026-02-04 (Estimated); Primary Completion 2031-02-04 (Estimated); Study Completion 2033-02-04 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 3 years
  Progression-free survival is calculated from the date of randomization to the date of documented local or regional relapse, distant metastasis, or death from any cause, whichever occurred first.

SECONDARY OUTCOMES:
Overall survival | 3 years
  Overall survival is calculated from the date of randomization to death from any cause.
Locoregional recurrence-free survival | 3 years
  Locoregional recurrence-free survival is calculated from the date of randomization to the date of documented locoregional recurrence or death from any cause.
Distant metastasis-free survival | 3 years
  Distant metastasis-free survival is calculated from the date of randomization to the date of documented distant metastasis or death from any cause.
Incidence of acute toxicity as assessed by CTCAE v5.0 | 3 years
  Acute adverse events (those that occurred within 1 year of randomisation) are graded according to the Common Terminology Criteria for Adverse Events (version 5.0).
Incidence of late toxicity as assessed by the Late Radiation Morbidity Scoring Scheme of the Radiation Therapy Oncology Group | 3 years
  Late adverse events (those occurring >1 year after randomisation) are graded according to the Late Radiation Morbidity Scoring Scheme of the Radiation Therapy Oncology Group.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China